CLINICAL TRIAL: NCT02962037
Title: Are Patients Suffering From DSPS Show Compromising in Everyday Functions and Abilities (Attention and Concentration, Mood and Fatigue) Before Handling the Disorder? And Whether the Treatment Fixes the Disorder?
Brief Title: Are Patients Suffering From DSPS Show Compromising in Everyday Functions and Abilities Before Handling the Disorder?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lilach Kemer (Other)
Responsible Party: Sponsor-Investigator, Lilach Kemer, Dr., Assuta Medical Center
Organization: Assuta Medical Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0092-16-ASMC
Record Dates: First submitted 2016-10-30; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Delayed Sleep Phase Syndrome
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Base line (No Intervention): the subject will take the tests in the morning and the evening
- After treatment (Experimental): the subject will take the tests in the morning and the evening
  Interventions: Other: Melatonin and light therapy

INTERVENTIONS:
Other: Melatonin and light therapy
  Arms: After treatment

SUMMARY:
The purpose of this study is to determine whether the known treatment for DSPS also improve the cognitive ability and mood of the patients.

DETAILED DESCRIPTION:
Every participant will take a few test and tasks that are going to test his cognitive ability and mood before treatment in 08:00 and 20:00, and again the same tests at the same hours after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with DSPS

Exclusion Criteria:

* attention deficit hyperactivity disorder - diagnosed, affective disorder- diagnosed

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Sleep patterns | 1 week
  Sleep actigraph
Melatonin secretion | 12 hours
  Melatonin -Sulfate Urine
Brief Symptom Inventory | 1 day
  BSI Questionnaire- assess the subject's emotional state
Epworth Sleepiness Scale | 1 day
  ESS Questionnaire- measure daytime sleepiness
Karolinska Sleepiness Scale | 1 day
  KSS Questionnaire- self-reported, subjective assessment of the subject's level of drowsiness
Continuous Performance Test 3 | 1 day
  Task-oriented computerized assessment of attention-related problems

IPD SHARING:
Plan to Share IPD: No